CLINICAL TRIAL: NCT00897234
Title: Plasma Quantification of Cathepsin D and FAS in Non-Small Cell Lung Cancer
Brief Title: Blood Samples From Patients With Non-Small Cell Lung Cancer and From Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2008NTLS094; 0809M47482 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collection, one 10 ml purple top EDTA tube, will be collected from each patient and control via venipuncture or from a central line.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Volunteers: Non-smoking healthy volunteers
  Interventions: Other: Mass Spectrometry
- Non-Small Cell Lung Cancer: Patients with non-small cell lung cancer.
  Interventions: Other: Mass Spectrometry

INTERVENTIONS:
Other: Mass Spectrometry — Levels of Cathepsin D (CD) and fatty acid synthase (FAS) will be measured using isobaric tag labeling coupled with mass spectrometry. RNA concentration will be measured using spectrophometer and purity will be analyzed.

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at blood samples from patients with non-small cell lung cancer and from healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Measure plasma cathepsin D levels in patients with non-small cell lung cancer and in healthy volunteers using mass spectometry.
* Measure fatty acid synthase levels in these patients and healthy volunteers using mass spectometry.

OUTLINE: Blood samples are collected from patients and healthy volunteers to measure the levels of cathepsin D and fatty acid synthase by proteomic profiling and mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

Non-Small Cell Lung Cancer Patients

* Documented diagnosis of non-small cell lung cancer, any stage and any time point in the course of treatment (i.e., at diagnosis, during any treatment, and during post treatment surveillance)
* Measurable disease by CT scan within the past 4 weeks

Healthy volunteer

* Non-smoking, defined as < 5 packs/year history of smoking and cessation of smoking ≥ 6 months ago OR a never smoker

  * Not regularly exposed (i.e., daily) to second-hand smoke

Exclusion Criteria:

* Severe underlying lung disease (i.e., chronic obstructive pulmonary disease with FEV_1 < 1.0 L, pulmonary fibrosis, bronchiectasis, cystic fibrosis, etc.) as determined by enrolling researcher.

Written consent must be given for both subjects and controls.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have non-small cell lung cancer (NSCLC) will be recruited from the Masonic Cancer Center at the University of Minnesota. Controls will be non-smoking individuals, age matched to the NSCLC subjects recruited through advertising. Normal controls should not be regularly exposed to second hand smoke.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Levels of cathepsin D | At Routine Follow-Up
  Measure plasma CD levels in patients with non-small cell lung cancer and non-smoker healthy controls using mass spectrometry.

SECONDARY OUTCOMES:
Levels of fatty acid synthase (FAS) | At Routine Follow-Up
  Measure FAS levels in patients with non-small cell lung cancer and non-smoker healthy controls using mass spectrometry.
Global microRNA expression | At Routine Follow-Up
  Measure global microRNA expression by microarray analysis using Illumina probes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Kratzke, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States